CLINICAL TRIAL: NCT02913690
Title: Effects of Dietary Supplementation Using Palm Tocotrienols in Chronic Hemodialysis (PATCH) Patients - A Multicenter Study Evaluating Markers of Inflammation, Oxidative Stress and Blood Lipids
Brief Title: Palm Tocotrienols in Chronic Hemodialysis (Malaysia) (PATCH)
Acronym: PATCH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Wayne State University (Other)
Collaborators: Universiti Putra Malaysia (Other); Malaysia Palm Oil Board (Other Government); PEMANDU (Unknown); National Kidney Foundation, United States (Other); Ministry of Health, Malaysia (Other Government)
Responsible Party: Principal Investigator, Associate Professor Dr Tilakavati Karupaiah, Associate Professor, National University of Malaysia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN-041-2015; NMRR-14-1859-23386 (Other: Medical Research and Ethics Committee)
Record Dates: First submitted 2016-04-26; First posted 2016-09-26 (Estimated); Last update posted 2020-05-21 (Actual); Status verified 2020-05

CONDITIONS: Chronic Kidney Failure
Keywords: Hemodialysis; Tocotrienol; Vitamin E
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Vitamin E

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator): Control group will be supplemented with placebo for 12 months.
  Interventions: Dietary Supplement: Placebo
- Intervention group (Active Comparator): The intervention arm will be supplemented with TRF for 12 months.
  Interventions: Dietary Supplement: TRF

INTERVENTIONS:
Dietary Supplement: Placebo — 2 x 150mg capsules daily
  Arms: Control group
Dietary Supplement: TRF — 2 x 150mg capsules daily
  Other Names: Vitamin E
  Arms: Intervention group

SUMMARY:
This study aims to determine if tocotrienol rich fraction (TRF) supplementation can improve markers of inflammation, oxidative stress and blood lipids in Malaysian hemodialysis (HD) patients.

DETAILED DESCRIPTION:
This study is a multi-centered, randomized, double blind, placebo-controlled trial where a total of 400 HD patients (200 supplemented; 200 control) will be recruited from government and private settings. Subjects will be randomized to either the intervention or control group. The intervention group will receive TRF (300 mg), daily for 12 months while the control group will only receive placebo, daily for 12 months. In addition, both groups will receive standard dietary counseling to ensure compliance to medical nutrition therapy guidelines for dialysis patients.

Patients who consented will be first subjected to a screening for identification of eligible subjects. The screening will involve basic anthropometry measures (height, weight, BMI), routine biochemistry result obtained from medical record, assessment of nutritional status and dietary evaluation. About 15ml of pre-dialysis blood will be collected by respective nurses for additional laboratory parameters (hsCRP, atherogenic profile and other inflammatory markers).

Patients who fulfill the inclusion criteria will be randomized to either control or intervention group. During the 12 months of treatment period, patients in both control and intervention groups will be assessed at baseline and 3-monthly intervals for laboratory results, medical condition, hospitalizations, nutritional status, dietary intake and compliance towards supplementation (intervention group only). A final measurement will be taken 3 months after study completion as a post follow up assessment upon cessation of supplementation. In all, patient data will be generated at 6 time points.

(A similar study, following a similar protocol and using the same study design and intervention will recruit 400 patients total (200 for each group) in Michigan, USA).

ELIGIBILITY:
Inclusion Criteria:

* Provided consent and comply to study protocol
* Undergoing HD treatment thrice-weekly for > 3 months
* Adequately dialyzed (Kt/V> 1.2 or urea reduction ratio (URR) of 65%) and hsCRP level <20 mg/dL.

Exclusion Criteria:

* Participated in another clinical trial involving an investigational product in the past 12 weeks preceding enrolment.
* Planned for kidney transplant over the study duration.
* Intake of vitamin E-containing supplements (>60 IU/day) 30 days preceding enrolment.
* Intake of anti-inflammatory medication except aspirin <325 mg/day in the past 30 days preceding enrollment.
* Female patients who are pregnant, lactating or planning a pregnancy during the course of the trial.
* Poor adherence to HD or medical treatment
* Patient with temporary catheter for dialysis access at baseline, or patients receiving graft/fistula within the 6-month study period.
* History of hospitalizations (>2 times within the past 90 days or one hospitalization within the 30 days) preceding enrollment.
* Receiving nutritional support ( via enteral and intra-venous route).
* Diagnosed with HIV/AIDS and/or on the anti-HIV therapy
* Receiving active treatment for cancer (excluding basal cell carcinoma of the skin).
* Patients with Hepatitis B or C.
* Any other significant disease or disorder where in the opinion of the respective nephrologist may affect the end results of this study
* Patients with a known allergy towards fish.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 336 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-12-14 (Estimated)

PRIMARY OUTCOMES:
Improvement in inflammatory marker based on the mean change from baseline to 12 months. | Baseline to 12 months
  Changes in biochemistry marker namely hsCRP (mg/dL)

SECONDARY OUTCOMES:
Changes in plasma lipids | Baseline to 12 months
  Based on biochemistry results for TC, LDL-C, HDL-C, triglyceride (TG), atherogenic profile, cholesteryl ester transfer protein (CETP), lecithin cholesterol acyltransferase (LCAT), apolipoprotein A1(ApoA1), apolipoprotein B-100 (ApoB-100)
Changes in restless leg syndrome scoring | Baseline to 12 months
  Based on restless leg syndrome questionnaire
Changes in anthropometry measures | Baseline to 12 months
  This includes body mass index (kg/m2) and skin fold measurements such as mid arm circumference (cm), mid-arm muscle circumference (cm), mid-arm muscle area (cm2) and triceps skin fold (mm)
Changes in body composition | Baseline to 12 months
  Body composition assessment pertaining to hydration status, lean tissue mass and fat mass is derived using a portable BIA device.
Changes in muscle strength | Baseline to 12 months
  Handgrip strength (in kilogram) will be measured using hand held dynamometer
Changes in biochemistry parameters | Baseline to 12 months
  Routine blood parameters (renal, liver function,lipid, hematology profile and dialysis adequacy) will be obtained from patients' medical records. Additional fasted blood sampling will be obtained to determine lipid biomarkers (CETP, LCAT, ApoA1, ApoB-100, lipoprotein particles) as well as inflammation and oxidative stress markers (hs-CRP, IL-6, F-isoprostane).
Changes in dietary intake | Baseline to 12 months
  Dietary intake will be assessed using a 3-day 24-hr diet recalls to determine macro and micronutrient intake.
Changes in nutritional status | Baseline to 12 months
  Patients will be screened with the Malnutrition Inflammation Score questionnaire to categorize their nutritional status.
Changes in qualify of life (QOL) | Baseline to 12 months
  Subjects will be interviewed using SF-36 & KD-QOL questionnaire which will derive QOL score.
Changes in rate of hospitalisation | Baseline to 12 months
  Difference in frequency of hospitalisation between the groups during the 12 months will be determined.
Changes in metabolomics analyses | Baseline to 12 months
  Metabolomic analyses (using blood specimens) will be carried out to determine differences in metabolites between the groups.

CONTACTS AND LOCATIONS:
Overall Officials: Tilakavati Karupaiah, PhD, Principal Investigator — National University of Malaysia
Locations (4):
- Malaysia (4):
  - UKM Medical Centre, Kuala Lumpur, Cheras
  - Hospital Serdang, Kajang, Selangor
  - National Kidney Foundation (Malaysia), Petaling Jaya, Selangor
  - Hospital Kuala Lumpur, Kuala Lumpur

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Daud ZA, Tubie B, Sheyman M, Osia R, Adams J, Tubie S, Khosla P. Vitamin E tocotrienol supplementation improves lipid profiles in chronic hemodialysis patients. Vasc Health Risk Manag. 2013;9:747-61. doi: 10.2147/VHRM.S51710. Epub 2013 Nov 28. PMID 24348043
- [Background] Boaz M, Smetana S, Weinstein T, Matas Z, Gafter U, Iaina A, Knecht A, Weissgarten Y, Brunner D, Fainaru M, Green MS. Secondary prevention with antioxidants of cardiovascular disease in endstage renal disease (SPACE): randomised placebo-controlled trial. Lancet. 2000 Oct 7;356(9237):1213-8. doi: 10.1016/s0140-6736(00)02783-5. PMID 11072938
- [Background] Locatelli F, Fouque D, Heimburger O, Drueke TB, Cannata-Andia JB, Horl WH, Ritz E. Nutritional status in dialysis patients: a European consensus. Nephrol Dial Transplant. 2002 Apr;17(4):563-72. doi: 10.1093/ndt/17.4.563. PMID 11917047
- [Background] Sagheb MM, Dormanesh B, Fallahzadeh MK, Akbari H, Sohrabi Nazari S, Heydari ST, Behzadi S. Efficacy of vitamins C, E, and their combination for treatment of restless legs syndrome in hemodialysis patients: a randomized, double-blind, placebo-controlled trial. Sleep Med. 2012 May;13(5):542-5. doi: 10.1016/j.sleep.2011.11.010. Epub 2012 Feb 7. PMID 22317944
- See also: Information on the parallel study conducted in USA by Wayne State University — https://clinicaltrials.gov/ct2/show/NCT02358967?term=patch+tocotrIENOL&rank=1